CLINICAL TRIAL: NCT02487329
Title: Efficacy of Er,Cr:YSGG Laser Irradiation Combined With Resin Based Tricalcium Silicate and Calcium Hydroxide on Direct Pulp Capping: a Randomized Clinical Trial
Brief Title: The Effect of Laser Combined With Pulp-capping Agents on Direct Pulp Capping
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Near East University, Turkey (Other)
Responsible Party: Principal Investigator, Esra Cengiz, DDS,PhD, Near East University, Turkey
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2015/30-197
Record Dates: First submitted 2015-06-22; First posted 2015-07-01 (Estimated); Last update posted 2015-07-01 (Estimated); Status verified 2015-06

CONDITIONS: Dental Pulp Exposure
Keywords: Direct pulp capping; Er,Cr:YSGG laser; Tricalcium silicate
MeSH Terms: conditions — Dental Pulp Exposure | interventions — Calcium Hydroxide; Dycal; CMW cement

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Calcium hydroxide (Active Comparator): Direct pulp capping with a self-hardening calcium hydroxide paste
  Interventions: Other: Calcium Hydroxide
- Er,Cr:YSGG laser + calcium hydroxide (Experimental): Direct pulp capping using Er,Cr:YSGG laser combined with calcium hydroxide
  Interventions: Other: Er,Cr:YSGG laser + calcium hydroxide
- TheraCal LC (Experimental): Direct pulp capping with resin based tricalcium silicate material
  Interventions: Other: TheraCal LC
- Er,Cr:YSGG laser + TheraCal LC (Experimental): Direct pulp capping using Er,Cr:YSGG laser combined with resin based tricalcium silicate material
  Interventions: Other: Er,Cr:YSGG laser + TheraCal LC

INTERVENTIONS:
Other: Calcium Hydroxide — Exposed area was sealed with a self-hardening calcium hydroxide paste then final restoration was completed using a resin-modified glass ionomer and a nanohybrid composite resin
  Other Names: Dycal, Dentsply, Tulsa, OK, USA
  Arms: Calcium hydroxide
Other: Er,Cr:YSGG laser + calcium hydroxide — After the exposed area was irradiated with Er,Cr:YSGG laser at an energy level of 0,5 W, a repetition rate of 20 Hz, 140 µs pulse duration with 0% water and 45% air for 10 s, it was sealed with a self-hardening calcium hydroxide paste.Then final restoration was completed using a resin-modified glass ionomer and a nanohybrid composite resin
  Other Names: Er,Cr:YSGG laser (Waterlase MD, Biolase, Irvine, CA, USA)
  Arms: Er,Cr:YSGG laser + calcium hydroxide
Other: TheraCal LC — TheraCal LC was applied directly to the exposed pulp with a needle tip syringe in incremental layers that was not to exceed 1 mm in depth. Then final restoration was completed using a resin-modified glass ionomer and a nanohybrid composite resin
  Other Names: TheraCal LC, Bisco, Schaumburg, Illinois, USA
  Arms: TheraCal LC
Other: Er,Cr:YSGG laser + TheraCal LC — After the exposed area was irradiated with Er,Cr:YSGG laser at an energy level of 0,5 W, a repetition rate of 20 Hz, 140 µs pulse duration with 0% water and 45% air for 10 s, TheraCal LC was used to seal the treated area. Then final restoration was completed using a resin-modified glass ionomer and a nanohybrid composite resin
  Arms: Er,Cr:YSGG laser + TheraCal LC

SUMMARY:
The purpose of this randomized clinical study was to evaluate the efficiency of Er,Cr:YSGG laser irradiation combined with a resin based tricalcium silicate material and calcium hydroxide (CH) in direct pulp capping for 3 months follow-up period.Sixty permanent vital teeth without symptoms and radiographic changes were randomly assigned to 4 groups (n=15): Gr 1: The exposed area was sealed with CH paste, Gr 2: The treated area was sealed with CH paste following Er,Cr:YSGG laser irradiation at an energy level of 0,5 W without water and 45% air, Gr 3: Resin based tricalcium silicate material (TheraCal LC) was applied directly to the exposed pulp, Gr 4: TheraCal LC was applied following irradiation with Er,Cr:YSGG laser.

DETAILED DESCRIPTION:
CH is used as gold standard in pulp capping procedures due to its beneficial properties such as induction of mineralization and inhibition of bacterial growth; however tunnel defects and cell inclusions in dentin bridges formed by CH may lead to leakage and bacteria penetration resulting in loss of vitality.

TheraCal LC is a new light-cured, resin-modified, tricalcium silicate based material designed to use for direct and indirect pulp-capping aiming to achieve a bond to composite resins thus reducing micro-leakage.The formulation of TheraCal LC containing tricalcium silicate particles in a hydrophilic monomer provides significant calcium release that stimulates hydroxyapatite and secondary dentin bridge formation The use of laser for direct pulp capping has been suggested for the considerable advantages of lasers including decontamination effect, biostimulation effect, hemostatic and coagulant effect.The erbium, chromium-doped:yttrium, scandium, gallium and garnet (Er,Cr:YSGG) laser which is a relatively new device has been reported to ablate dental hard tissues thanks to its high absorption in water and also strong absorption by the hydroxyl radicals present in the hydroxyapatite structure

ELIGIBILITY:
Inclusion Criteria:

* Permanent teeth with deep caries without symptoms
* Vital teeth
* No periapical radiographic changes
* The diameter of the exposed area is between 0,5 mm to 1,5 mm

Exclusion Criteria:

* Spontaneous pain,
* Tenderness to percussion and palpation,
* Bleeding lasting over 3 minute after exposure,
* Periapical radiographic changes such as periradicular or furcal radiolucency, a widened periodontal ligament space and resorption.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-01; Primary Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Pulp vitality | 3 months
  Pulp vitality is assessed with electric pulp tester as vital or non-vital
Assessment of pain with questionnaire | 3 months
  Pain assessment is carried out using the pain Numerical Rating Scale (NRS) with ratings between 0 to 9. No reactions to thermal stimuli and no tenderness to percussion.

SECONDARY OUTCOMES:
Radiographic success | 3 months
  No signs of root resorption (internal or external), no signs of furcation involvement or periapical radiolucency, no signs of loss of lamina dura, no widened periodontal ligament space

CONTACTS AND LOCATIONS:
Overall Officials: Hasan Guney Yılmaz, DDS,PhD, Study Director — Near East University

REFERENCES:
- [Result] Olivi G, Genovese MD, Maturo P, Docimo R. Pulp capping: advantages of using laser technology. Eur J Paediatr Dent. 2007 Jun;8(2):89-95. PMID 17571933
- [Result] Yazdanfar I, Gutknecht N, Franzen R. Effects of diode laser on direct pulp capping treatment : a pilot study. Lasers Med Sci. 2015 May;30(4):1237-43. doi: 10.1007/s10103-014-1574-8. Epub 2014 Apr 23. PMID 24756324